CLINICAL TRIAL: NCT01692210
Title: The Effect of Dexmedetomidine on Immunological Parameters of Women Undergoing Breast Cancer Surgery
Brief Title: The Effect of Dexmedetomidine of the Immune System
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: PA12-0524
Record Dates: First submitted 2012-09-19; First posted 2012-09-25 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Dexmedetomidine; Unilateral mastectomy; Blood sample collections; Immune system; White blood cell levels
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 15cc of blood drawn prior or at the moment of anesthesia induction and the morning after surgery.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Blood Draw Pre and Post Surgery: Patients within the UT MD Anderson Cancer Center who are scheduled for breast cancer surgery.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — After induction of general anesthesia, a loading dose of dexmedetomidine (1 mcg/kg) given in 15 min followed by an infusion of the same medication at a rate of 0.4 - 0.7 mcg/kg/hour.

SUMMARY:
The goal of this research study is to learn about how dexmedetomidine (a standard of care sedative) affects your immune system (your defenses against cancer) by measuring your white blood cell levels before and after surgery.

DETAILED DESCRIPTION:
Dexmedetomidine is a type of sedative used as part of anesthetic care. It is sometimes used to help lower the amount of pain killers and other anesthetics that are given to a patient during surgery. Researchers want to study how this drug works in cancer patients and review the patient's chart for pain levels and medication use after surgery. Part of this research involves studying the immune system of surgery patients.

If you agree to take part in this study, blood (about 1 tablespoon) will be drawn before you have surgery and the morning after surgery while you are still in the hospital. This blood will be used to learn more about how your immune system works.

After your second blood draw, your participation in this study will be over.

This is an investigational study.

Up to 20 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 - Women undergoing unilateral mastectomy for malignancy at MD Anderson Cancer Center.

3.1.2 - Patients 18 years of age and older. There will be no upper age restriction.

3.1.3 - Patients must sign a study-specific consent form.

Exclusion Criteria:

3.2.1 - ASA 4

3.2.2 - Contraindication to the use of dexmedetomidine.

3.2.2.1. Decompensated congestive heart failure.

3.2.2.2. Second and third degree heart block.

3.2.2.2. Known allergy to dexmedetomidine or any of the medications used in the study

3.2.3 - Patients taking clonidine for treatment of arterial hypertension.

3.2.4 - Patients that are pregnant.

3.2.5 - Patients taking opioids at the time of surgery.

3.2.6 - Patients having plastic surgical reconstruction.

3.2.7 - Recent chemotherapy (< 4 weeks).

3.2.8 - Active autoimmune or immunological disease including but not limited to systemic lupus erythematous, rheumatoid arthritis and Sjogren's disease

3.2.9 - Patient refusal to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing unilateral mastectomy for malignancy at MD Anderson Cancer Center in Houston, Texas.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pre and Post Surgical Lymphocyte Counts | 2 days
  Lymphocyte counts determined by flow-cytometry and their function by cytotoxicity assays performed in the laboratory using samples obtained before and the morning after surgery. Patients who experience a reduction of less than 50% of their preoperative natural killer cell (NKC) activity considered as a success.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P. Cata, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org